CLINICAL TRIAL: NCT04954105
Title: Influence of the COvid-19 Epidemic on STRESS and Heart-Rate Variability in Health-care Workers
Acronym: COVISTRESS HRV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital of Clermont-Ferrand (CHU), Clermont-Ferrand, France (Unknown); UMR CNRS 6024 LaPSCo, Clermont-Ferrand, France (Unknown); Wittyfit, Paris, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020 COVISTRESS HRV
Record Dates: First submitted 2021-07-06; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Stress; Heart Rate Variability, Biomarker of Stress; Burnout
Keywords: Stress; Coronavirus; HAZMAT; Epidemics
MeSH Terms: conditions — Burnout, Psychological; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COVID-19 pandemic is an exceptional and particularly anxiety-provoking health situation. In particular, for healthcare professionals who come into contact with patients who are contaminated or suspected of contamination, such as emergency rooms. The management of these patients requires reinforced protective equipment. However, in the context of this pandemic, data is currently non-existent on the objective measurement of the stress of these professionals. Sinus variability of heart rate is a biomarker of stress measured with a simple heart rate monitor or a watch, completely painless, non-intrusive, and used by the general public routinely in many areas (monitoring sports sessions, etc.).

DETAILED DESCRIPTION:
This is an observational study. In the emergency room, each participant will wear a heart rate monitor and a consumer watch throughout the working day (there will be no measurement on duty at night, nor measurement at home). The days will be notified as being in the "COVID sector", "non-COVID sector" or "Trauma Room".

Each participant will complete a questionnaire comprising visual analog scales on the feeling (health concern, stress, fatigue, quality of sleep, anxiety, morale, burnout, decisional latitude, psychological demand, support, self-esteem), time of start and end of work, and socio-demographic data (sex, age, weight, height, smoking)

ELIGIBILITY:
Inclusion Criteria:

* Emergency health care worker

Exclusion Criteria:

* refusal to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Emergency health care worker
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Heart-Rate Variability (HRV) | up to day 1
  HRV is a measure of the variation in time between each heartbeat. This variation is controlled by the autonomic nervous system. It works regardless of our desire and regulates, among other things, our heart rate, blood pressure, breathing, and digestion. It will be assess by heart rate monitor

SECONDARY OUTCOMES:
Stress | hours 0 at day 1
  Stress level will be assessed by questionnaire
Stress | hours 24 at day 1
  Stress level will be assessed by questionnaire
Perception of the epidemic | day 1
  Perception of the epidemic will be assessed by questionnaire
Sociodemographic factors and lifestyle habits | day 1
  Sociodemographic factors and lifestyle habits will be assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Bouillon-Minois, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France